CLINICAL TRIAL: NCT06879119
Title: Clinical Efficacy Study of Localized Scalp Thread Embedding in the Treatment of Male Androgenetic Alopecia
Brief Title: Clinical Evaluation of Localized Scalp Thread Embedding for Male Androgenetic Alopecia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing University of Chinese Medicine, Shenzhen Hospital (Other)
Responsible Party: Principal Investigator, Aijuan Wang, Attending Physician, M.D., Beijing University of Chinese Medicine, Shenzhen Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JDF-IRB-2021050102
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Androgenetic Alopecia
Keywords: Androgenetic Alopecia; Interventional study; Non-pharmacological interventions
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Observational cohort: localized scalp thread embedding (Other): All participants meeting the inclusion criteria underwent a standardized scalp thread embedding procedure targeting the vertex alopecic area. Participants were prospectively observed for 6 months, with monthly follow-up assessments to evaluate outcomes . No additional interventions were administered during follow-up.
  Interventions: Procedure: Localized scalp thread embedding

INTERVENTIONS:
Procedure: Localized scalp thread embedding — Volunteers who met the inclusion criteria were enrolled in the trial. All participants underwent treatment intervention in the vertex alopecic area via vertex alopecic area scalp thread embedding. A single thread embedding session was performed upon enrollment, with monthly follow-ups conducted over a total period of 6 months. Operative procedure: After fully exposing and disinfecting the treatment area, threads were inserted into the scalp at an approximately 15-degree oblique angle, with needle tips reaching the subgaleal space at a depth of 2-4 mm. Threads were spaced 1 cm apart. Upon completion, the treated area was disinfected and applied with erythromycin ointment.

SUMMARY:
This clinical study aims to evaluate a breakthrough treatment for hair loss (androgenetic alopecia, AGA) using dissolvable threads placed under the scalp skin. The investigators hypothesize that these specially designed threads can improve hair growth, avoiding the need for invasive surgery.

Current AGA treatments taken orally often have limitations, prompting researchers to explore localized approaches. While early studies show promise for localized scalp thread embedding, three key challenges remain: 1) No standardized way to measure effectiveness, 2) Lack of objective biological markers to track progress, and 3) Limited understanding of how exactly these treatments work.

This study addresses these gaps through precise thread placement in balding areas, following international dermatology guidelines. Using advanced measurement tools, the investigators will track changes in hair thickness (primary measure), blood flow patterns under the skin, and oil gland activity (secondary measures). By focusing on one key treatment factor, this research provides the first comprehensive evidence showing how this minimally invasive approach may slow or reverse AGA progression.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Age 18-50 years
* No clinically significant comorbidities
* Androgenetic alopecia (Hamilton-Norwood III-V)
* No systemic anti-hair loss therapy use within 3 months
* No topical hair regrowth agent use within 3 months

Exclusion Criteria:

* Active scalp infection
* Scalp psoriasis
* Scalp eczema
* Open scalp wounds
* Allergy to thread materials
* Uncontrolled diabetes mellitus
* Immunodeficiency disorders
* Non-compliance with follow-up visits
* Refusal to provide informed consent
* Investigator-deemed contraindications

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
Hair Shaft Parameters | From enrollment to the end of treatment at 6 months
  The German FotoFinder trichoscopy system (FotoFinder Systems GmbH, Birbach, Germany) was utilized, incorporating its integrated trichometric analysis module and high-resolution optical imaging system (Medicam 1000HD) with 20X-140X magnification. Hair shaft parameters include: total hair count, hair density, hair shaft diameter, and hair follicle typing.

SECONDARY OUTCOMES:
Scalp thickness | From enrollment to the end of treatment at 6 months
  Scalp thickness measured by B-mode ultrasound（Acuson S1000，Siemens AG，Germany）
Scalp blood flow | From enrollment to the end of treatment at 6 months
  Scalp blood flow velocity assessed by Doppler ultrasound （Acuson S1000，Siemens AG，Germany）
Scalp sebum production | From enrollment to the end of treatment at 6 months
  The scalp sebum measurement was performed using the German Sebumeter SM815 (Courage & Khazaka electronic GmbH, Germany), with sebum test kits procured from Beijing Jinhongfan Trading Co., Ltd. The quantification principle adheres to the internationally recognized SEBUMETER® methodology, which employs photometric analysis to quantify sebum content by measuring light transmittance through a 0.1-mm-thick matte-finish adhesive film that absorbs cutaneous lipids.

CONTACTS AND LOCATIONS:
Locations (1):
- Dongfang Hospital Beijing University of Chinese Medicine, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No